CLINICAL TRIAL: NCT05559151
Title: Effect and Mechanism of Remimazolam Benzenesulfonate on Eenhanced Recovery After Surgery in Patients Undergoing Radical Gastrectomy for Gastric Cancer
Brief Title: Effect and Mechanism of Remimazolam Benzenesulfonate on Enhanced Recovery After Surgery in Patients Undergoing Radical Gastrectomy for Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhonghua Chen,MD (Other)
Collaborators: China (Zhejiang) Health technology RESEARCH and development and transformation platform (Unknown)
Responsible Party: Sponsor-Investigator, Zhonghua Chen,MD, associate chief physician, Shaoxing Hospital of Zhejiang University
Organization: Shaoxing Hospital of Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IEC-K-AF-074-1.0
Record Dates: First submitted 2022-09-25; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Remimazolam Benzenesulfonate on Nenhanced Recovery After Surgery; Possible Molecular Mechanism of Remimazolam Benzenesulfonate
Keywords: Remimazolam Benzenesulfonate; ERAS; Radical Gastrectomy for Gastric Cancer

STUDY DESIGN:
Intervention Model Description: Sixty patients undergoing radical gastrectomy for gastric cancer were selected and divided into two groups according to random number table method: control group (group P) and experimental group (group R), with 30 cases in each group. All enrolled patients signed informed consent. Control group: the control group (group P) received target controlled infusion of propofol. Experimental group: the experimental group (group R) received target controlled infusion of remimazolam benzenesulfonate. And the BIS value of the two groups was controlled at 50±5.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the experimenters nor the participants knew whether they were getting an experimental drug or a placebo. In this way, the description of the therapeutic effects and adverse reactions of the subjects, as well as the record of the various reactions of the experimenters, can be as objective as possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (group R) (Experimental): The experimental group (group R) received target controlled infusion of remimazolam benzenesulfonate, and the BIS value was controlled at 50±5.
  Interventions: Procedure: Remimazolam Benzenesulfonate
- the control group (group P) (Placebo Comparator): the control group (group P) received target controlled infusion of propofol, and the BIS value was controlled at 50±5.
  Interventions: Procedure: Remimazolam Benzenesulfonate

INTERVENTIONS:
Procedure: Remimazolam Benzenesulfonate — In the experimental group, remazolam 6-12mg/kg/h, atracurium cisphenylate 0.1-0.3 mg/kg and sufentanil 0.3-0.5 μg/kg were infused by micropump for anesthesia induction, and the BIS value was controlled at 50±5 before tracheal intubation.
  Anesthesia maintenance: intravenous infusion of remifentanil 0.1-0.3 μg/kg/min, target controlled infusion of remifentanil in experimental group (group R), BIS value was controlled at 50±5, intermittent addition of atracurium cisphenylate to maintain muscle relaxation.

SUMMARY:
The purpose of this study is to discuss the benzene sulfonic acid red horse azole shimron the occurrence of postoperative complications in patients with gastric cancer radical and its severity, at the same time, comparing the control group (propofol) the degree of inflammation in patients with different time points difference, preliminary in this paper, the benzene sulfonic acid red horse azole shimron in gastric cancer radical viscera molecular mechanism of protection and quick recovery.

DETAILED DESCRIPTION:
A total of 60 patients undergoing radical gastrectomy for gastric cancer were randomly divided into control group (group P) and experimental group (group R), with 30 cases in each group. Two groups are made by way of BIS target controlled infusion of anesthesia, experimental group (R group) target controlled infusion red horse azole shimron, control group (P group) target controlled infusion of propofol, BIS values are controlled in 50 + 5, postoperative observation of dynamic changes of inflammatory cytokines in plasma, postoperative adverse reactions, postoperative recovery, postoperative 30-day mortality and postoperative complications.

Through statistical analysis, it is proposed that remazolam can stabilize perioperative hemodynamic fluctuation, improve postoperative recovery, reduce the release of inflammatory mediators, reduce complications, shorten the length of hospital stay, reduce hospitalization costs, and accelerate the rapid recovery of patients with radical gastrectomy. It is proved that remazolam besylate can reduce the inflammatory response of patients undergoing radical gastrectomy, reduce the incidence of postoperative complications, and provide a favorable supplement to ERAS in patients undergoing radical gastrectomy. At the same time provide more red horse azole shimron, applied to the systemic narcotic induction and maintenance of cases and further added red horse azole shimron applied to clinical usage and dosage (by age, gender, race, obesity status, ASA grade and weight the effect of covariate), adverse reactions, and other commonly used anesthetic synergy.

ELIGIBILITY:
Inclusion Criteria: Sixty patients undergoing elective laparoscopic radical gastrectomy for gastric cancer; aged 18-75 years; ASA≤ⅲ .

-

Exclusion Criteria: Emergency surgery or non-radical gastrectomy patients; age < 18 or > 75 years old, ASA grade ≥IV. Benzodiazepines or other narcotic drug allergy patients; patients with neurological and psychiatric disorders, long-term use of sedatives or antidepressants; has a history of alcoholism or drug dependence; intraoperative find distant metastasis; receive radiation and chemotherapy, cachexia; patients with a history of other malignant tumors within five years; the patient refused to participate in the study.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic changes of inflammatory cytokines in plasma | Before induction, 2 hours after the start of surgery, immediately after the end of surgery, 24 hours after the end of surgery, and 72 hours after the end of surgery
  Dynamic changes of inflammatory cytokines in plasma
Postoperative adverse reactions | Within one week after surgery
  Nausea, vomiting, respiratory depression, irritability
Postoperative recovery | Within one week after surgery
  Postoperative resuscitation time, tracheal intubation extubation time, catheter removal time, nasogastric tube removal time, first fluid diet time, first exhaust time, first ambulation time
Postoperative complications | Within one week after surgery
  pulmonary infection, oxygenation injury, arrhythmia, bleeding, intestinal paralysis, incision infection, renal insufficiency, cognitive dysfunction, etc.
mortality rate | Within 30 days after surgery
  mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoxing People's Hospital, Shaoxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No